CLINICAL TRIAL: NCT01989221
Title: Sancuso® in Patients With Nausea and/or Vomiting From Gastroparesis: An Open Label Study.
Brief Title: Sancuso® for Gastroparesis: An Open Label Study.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21086
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Placebo followed by Sancuso (Other): Placebo at baseline for one week followed by Sancuso® (granisetron transdermal system) 3.1 mg/24 hours for two weeks
  Interventions: Drug: Sancuso®

INTERVENTIONS:
Drug: Sancuso® — Sancuso® (granisetron transdermal system) 3.1 mg/24 hours

SUMMARY:
The aim of this study is to determine the efficacy of Sancuso® (granisetron transdermal system) 3.1 mg/24 hours in improving symptoms of nausea and vomiting in patients with gastroparesis. This will be a prospective open-label study using Sancuso® to treat symptoms of nausea and/or vomiting in patients diagnosed with gastroparesis. Symptomatic patients with diabetic or idiopathic gastroparesis with nausea and/or vomiting will be enrolled. The Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD) will be used to capture the severity of symptoms, including nausea and vomiting, at baseline for one week. Patients will then be treated with Sancuso®. Patients will continue to fill out the GCSI-DD on a daily basis while undergoing treatment with Sancuso® for two weeks. To determine if Sancuso® treatment helps improve symptoms of nausea and vomiting, the symptoms at baseline will be compared to symptoms after the first week and the second week of treatment. Thirty patients diagnosed with gastroparesis (approximately 15 with diabetic and 15 with idiopathic gastroparesis) will be treated on an open label basis with Sancuso®. The goal of this study is to demonstrate the efficacy of Sancuso® in treating nausea and/or vomiting in gastroparesis patients. Safety information will also be collected regarding any adverse effects. If the results are encouraging, as we expect them to be based on personal experience, a larger double blind study would be appropriate.

DETAILED DESCRIPTION:
Objectives The aim of this study is determine the efficacy of Sancuso® in improving symptoms of nausea and vomiting in patients with gastroparesis.

The specific objectives of this study are to determine:

1. Determine the treatment response of Sancuso® in gastroparetic patients with nausea and/or vomiting.
2. Determine which specific symptoms of gastroparesis improve - nausea, vomiting, early satiety, abdominal distension, abdominal pain
3. To determine symptomatic responses in both diabetic and idiopathic gastroparesis
4. To determine the time course of symptom improvement (with Sancuso® for symptoms of gastroparesis;

The hypotheses to be tested include:

1. Sancuso® improves symptoms of gastroparesis.
2. Symptoms of nausea and vomiting improve to a greater degree than abdominal pain.
3. The beneficial response of Sancuso® is seen in both diabetic and idiopathic gastroparesis.
4. The symptom reduction occurs on days 3 after starting treatment and continues throughout the treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age Diagnosed gastroparesis patients with symptoms of gastroparesis for at least 3 months Symptoms of nausea and vomiting of at least moderate severity using the GCSI Prior history of delayed gastric emptying as determined by scintigraphy Gastroparesis from either diabetic or idiopathic etiologies Symptoms of nausea and vomiting that have not responded adequately to conventional antiemetic agents (Compazine®, Tigan®)

Exclusion Criteria:

* Post-surgical gastroparesis Prolonged QTc on EKG Prior intolerance to 5HT3 antagonists (ondansetron or granisetron) Known hypersensitivity to granisetron or to any of the components of the patch Current treatment with ondansetron or granisetron. Patients may stop these medications for one week to enter the study. Patients will not be allowed to take ondansetron or oral granisetron during the study.

Use of ketoconazole, a medications with known drug-drug interactions with granisetron Women known to be pregnant, as determined on enrollment by a urine pregnancy test Women of childbearing potential who do not agree to use a medically approved form of contraception Nursing mothers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry P Parkman, MD, Principal Investigator — Temple University Hospital
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: goal was 20 patients, 14 entered
Period: Overall Study
Arm/Group | Placebo Followed by Sancuso
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Followed by Sancuso: Placebo - Control for 1 week followed by Sancuso® (3.1 mg/24 hours) for 2 weeks
Arm/Group | Placebo Followed by Sancuso
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: GCSI-DD Total Composite Symptom Scores.
Description: The Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD) was used to capture the severity of symptoms during one week at baseline and two weeks of treatment with GTS. The GCSI-DD includes questions about severity of nausea, early satiety, postprandial fullness, upper abdominal pain, and overall symptoms. Patients rated their symptom severity on a scale of 0 (no symptom), 1 (mild), 2 (moderate), 3 (severe), and 4 (very severe) and recorded the number of vomiting episodes per day. A daily composite score was calculated as the average of the five symptom scores (not including overall symptom severity) with a cap of 4 vomiting episodes per day.
Time Frame: Three weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo Followed by Sancuso: Placebo - Control followed by Sancuso® (granisetron transdermal system) 3.1 mg/24 hours
Arm/Group | Placebo Followed by Sancuso
Number analyzed (Participants) | 14
score on a scale
  Baseline | 1.89 (0.15)
  Week 1 of Treatment | 1.57 (0.20)
  Week 2 of Treatment | 1.34 (0.21)
Statistical Analysis 1: Comparison: Placebo Followed by Sancuso; Test type: Superiority; p < 0.01, t-test, 2 sided — Threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 0.55, Standard Deviation 0.12 — Mean GCSI-DD scores during one week at baseline were compared to mean GCSI-DD scores during the second week of Sancuso treatment

2. Secondary Outcome: Total Gastrointestinal Nausea and Vomiting Symptom Index
Description: The Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD) was used to capture the severity of symptoms during one week at baseline and at two weeks of treatment with GTS. The GCSI-DD includes questions about severity of nausea, early satiety, postprandial fullness, upper abdominal pain, and overall symptoms. Patients rated their symptom severity on a scale of 0 (no symptom), 1 (mild), 2 (moderate), 3 (severe), and 4 (very severe) and recorded the number of vomiting episodes per day. A daily composite score was calculated as the average of the five symptom scores (not including overall symptom severity) with a cap of 4 vomiting episodes per day.
Time Frame: Three weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Followed by Sancuso
Number analyzed (Participants) | 14
score on a scale
  Baseline | 2.31 (0.17)
  Week 1 of Treatment | 1.69 (0.28)
  Week 2 of Treatment | 1.30 (0.27)
Statistical Analysis 1: Comparison: Placebo Followed by Sancuso; Test type: Other; p < 0.01, t-test, 2 sided — Threshold for statistical significance was p < 0.05; Mean Difference (Final Values) = 1.01, Standard Deviation 0.27 — Mean nausea and vomiting symptom scores during one week at baseline were compared to mean symptom scores during the second week of Sancuso treatment

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Sancuso: Sancuso (3.1mg/24 hours) for 2 weeks
Arm/Group | Sancuso
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 10/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sancuso (N=14)
Itching (Skin and subcutaneous tissue disorders) | 2 (2)
Redness at the patch site (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Poor Patch Adherence (Product Issues) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT01989221/Prot_SAP_000.pdf